CLINICAL TRIAL: NCT01165866
Title: Ondansetron Vs Metoclopramide in the Treatment of Vomiting in Gastroenteritis Patients: A Randomized Controlled Trial
Brief Title: Ondansetron Versus Metoclopramide in Treatment of Vomiting in Gastroenteritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Dr Khalid M. Al Ansari, Hamad Medical Corporation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 8031/08
Record Dates: First submitted 2010-07-18; First posted 2010-07-20 (Estimated); Last update posted 2010-10-26 (Estimated); Status verified 2010-10

CONDITIONS: Gastroenteritis
Keywords: Ondansetron; Metoclopramide; Gastroenteritis
MeSH Terms: conditions — Gastroenteritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment 1. (Active Comparator): Metoclopramide 0.3 mg/kg max 10 mg in burette and mixed with normal saline to make up 50 cc of medication and normal saline as a single intravenous dose. Complete blood count,serum electrolytes,renal function,HCO3 level will be requested.Oral fluid will be started thereafter and increased gradually until patient discharge.
  Interventions: Drug: Treatment 1. Metoclopramide
- Treatment2. (Other): Ondansetron 0.15 mg/kg max 4 mg in burette and mixed with normal saline to make up 50 cc of medication and normal saline to be given over 10 minutes,then patient will be kept NPO for one hour after completion of the anti emetic infusion and last episode of vomiting . Oral fluid will be started thereafter and increased gradually until fully tolerated and the patient is ready for discharge
  Interventions: Drug: Treatment 2 Ondansetron

INTERVENTIONS:
Drug: Treatment 1. Metoclopramide — metoclopramide 0.3mg/kg maximum dose 10mg will be added in the burette and mixed with normal saline to make up 50cc of medication for intravenous administration.
  Other Names: primpran
  Arms: Treatment 1.
Drug: Treatment 2 Ondansetron — Single dose of Ondansetron 0.15 mg/kg
  Other Names: Zofrane
  Arms: Treatment2.

SUMMARY:
Is intravenous metoclopramid as effective as intravenous ondansetron in the treatment of persistent vomiting in patients with acute gastroenteritis.

DETAILED DESCRIPTION:
In this study, we will compare the efficacy of a single intravenous dose of ondansetron versus intravenous metoclopramide in the treatment of persistent vomiting in simple gastroenteritis in a larger RCT.

PEC Al Saad is the main Pediatric Emergency Center in the state of Qatar with approximately 200,000 visits annually. It has a capacity of 42 observation beds providing most of the inpatient facilities except for intensive care monitoring. Patients admitted to the PEC are managed there for 48 hours or longer if needed, they are then transferred to Hamad General Hospital for further investigation and completion of their treatment. Hamad General Hospital is the main tertiary care hospital in Qatar with a capacity of around 100 pediatric beds.

All acute gastroenteritis patient between 1-14 years presenting to PEC Al Saad with diarrhea, persistent vomiting , fail oral rehydration and admitted to the observation unit for intravenous hydration will be eligible for the study.

Patients were excluded from the study if they had one or more of the following: Previous abdominal surgery,Suspicion of surgical abdominal,Bile stained vomitus,History of hepatic illness,Metabolic diseases, including diabetes mellitus and in-born error of metabolism,Children with shock or impending shock,Sever dehydration,Previous hypersensitivity or abnormal reaction to metoclopramide or ondansetron,Parenteral antiemetic treatment in the previous 24hrs or Seizure disorder

One group will receive a single IV dose of Ondansetron after enrollment and the second group will receive a single IV dose of Metoclopramide On arrival to the PEC, patients with simple gastroenteritis will be assessed by the pediatric specialist on-call, patients with persistent vomiting who fail ORS therapy will be admitted for observation and management as usual. The pediatric specialist in the observation room will take history, perform full physical examination and evaluate the degree of dehydration . Patients will be assessed for eligibility to the study based on the aforementioned inclusion criteria.

Guardians of eligible patients will be approached regarding the study, explaining the purpose and the treatment modalities, patients will be included after obtaining a verbal and written consent. Complete blood count, serum electrolytes, renal function, HCO3 level will be requested for all study patients upon recruitment.

The observation physician will complete the data collection sheet that will include the patient's demographics, physical examination, degree of dehydrations , number, amount and time of every vomiting and diarrhea episode and lab work results.

Intravenous Ondansetron and intravenous metoclopramide treatment will be prepared by a pharmacist, who will put each treatment in a sealed coded envelope A and B depending on the content (Ondansetron or Metoclopramide). The code of intervention package will be deposited with the pharmacist. The medical team in addition to the patients will be blinded to the content of the envelopes. There will be no detectable difference in the color or smell of the different solutions, the amount of medication will be determined by the weight of the patient (Ondansetron 0.15mg/kg maximum dose 4mg, Metoclopramide 0.3 mg/kg maximum dose 10mg), medication will be added in the buret and mixed with normal saline to make up 50cc of medication and normal saline for intravenous administration.

Patients will receive a single intravenous dose of the study medication after enrollment over 10 minutes and intravenous fluids will be started at the rate required based on the percentage of dehydration. Patients will be kept NPO for one hour after the completion of the antiemetic infusion and last episode of vomiting, oral fluids will be started thereafter and increased gradually until fully tolerated and the patient is ready for discharge. If vomiting recur NPO period will be extended for another half an hour from the last vomit and oral fluids will be tried gradually until the patient is fit for discharge. Vomiting and diarrhea episodes will be recorded by time and amount throughout admission.

Duration of IV fluid therapy needed, observed study medication side effects all will be recorded until the patient is ready for discharge if extra-pyramidal side effect are seen or suspected diphen hydramine 1 mg/kg (maximum dose 50mg/dose) will be given over 5 minutes and the patient will be observed until free of symptoms. Addition interventions such as antibiotics, antipyretics will be recorded as additional therapies.

The treating physician will discharge patients based on clinical grounds such as tolerating oral fluids, improve hydration status, absent of significant fluid loss through stool and free of major medication side effects. Patients found to be fit for discharge, will have date and time of discharge documented. In addition parents will be asked to give a number ,that represent their perception of their child's nausea symptoms and oral intake improvement on discharge, 0-100, 0 indicates no improvement and 100 back to base line.

Discharge Patients will be sent home on oral fluid therapy and BRAT diet. All patients will be followed up for 72 hours post discharge by a phone call daily.

ELIGIBILITY:
Inclusion Criteria:

* All acute gastroenteritis patient between 1-14 years presenting to PEC Al Saad with diarrhea, persistent vomiting , fail oral rehydration and admitted to the observation unit for intravenous hydration will be eligible for the study.

Exclusion Criteria:

1. Previous abdominal surgery
2. Suspicion of surgical abdominal
3. Bile stained vomitus
4. History of hepatic and renal illnesses
5. In-born error of metabolism
6. Children with shock or impending shock
7. Sever dehydration.
8. Previous hypersensitivity or abnormal reaction to metoclopramide or ondansetron
9. Antiemetic treatment within 48 hours prior to presentation.
10. Seizure disorder

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 170 (Actual)
Dates: Start 2008-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
is the proportion of patients with cessation of vomiting after study medication administration in each group. | one year

SECONDARY OUTCOMES:
Time to complete cessation of vomiting, time to successful oral therapy,length of hospital stay, parents perception of the child nausea symptom and oral tolerance on discharge and daily follow up for 3 days. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Khalid M Al-Ansari, FRCPC,FAAP, Principal Investigator — Hamad Medical Corporation ,Weill Cornell Medical College
Locations (1):
- Pediatric Emergency Centre, Al-Saad, Doha, Qatar

REFERENCES:
- [Derived] Al-Ansari K, Alomary S, Abdulateef H, Alshawagfa M, Kamal K. Metoclopramide versus ondansetron for the treatment of vomiting in children with acute gastroenteritis. J Pediatr Gastroenterol Nutr. 2011 Aug;53(2):156-60. doi: 10.1097/MPG.0b013e3182132d8d. PMID 21788756